CLINICAL TRIAL: NCT04728646
Title: Evaluation of Dextenza in Patients With Ocular Graft Vs Host Disease (GVHD) and Effect on Ocular Surface Disease Outcomes.
Brief Title: Evaluation of Dextenza in Patients With Ocular GVHD and Effects on Ocular Surface Disease Outcomes
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Due to difficulty enrolling subjects whom had not meet the inclusion criteria
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Principal Investigator, Reza Dana, MD, Professor, Director of Epidemiology for Ophthalmology, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2020P003125
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Graft Vs Host Disease
Keywords: graft vs Host disease; GVHD; Dextenza; eye; ocular surface disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — Calcium Dobesilate

STUDY DESIGN:
Intervention Model Description: Eyes of enrolled patients will be randomized to treatment arms in a 1:1 ratio (Dextenza insert:control insert). All study participants will receive the Dextenza insert in the lower puncta of one eye (treatment eye) and a standard dissolvable intracanalicular plug in the lower puncta of the fellow eye (control eye).
Who Masked: Participant
Masking Description: The randomization results will also be communicated to the treating physician, who will administer the Dextenza and control plug in the respective eyes while keeping the patient blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- DEXTENZA (dexamethasone ophthalmic insert) 0.4 mg, for intracanalicular use (Experimental): All patients will receive Dextenza insert in one eye and a regular dissolvable intracanalicular plug in the fellow-eye (randomized).
  Interventions: Drug: DEXTENZA (dexamethasone ophthalmic insert) 0.4 mg, for intracanalicular use
- Dissolvable intracanalicular plug (Other): All patients will receive Dextenza insert in one eye and a regular dissolvable intracanalicular plug in the fellow-eye (randomized).
  Interventions: Device: Regular dissolvable intracanalicular plug

INTERVENTIONS:
Drug: DEXTENZA (dexamethasone ophthalmic insert) 0.4 mg, for intracanalicular use — Inserted During Screening/Baseline: Day Zero in either the right or left eye (depending on randomization)
  Arms: DEXTENZA (dexamethasone ophthalmic insert) 0.4 mg, for intracanalicular use
Device: Regular dissolvable intracanalicular plug — Inserted During Screening/Baseline: Day Zero in either the right or left eye (depending on randomization)
  Arms: Dissolvable intracanalicular plug

SUMMARY:
To evaluate the safety and efficacy of Dextenza intracanalicular insert in patients with ocular graft-versus-host disease (GVHD).

DETAILED DESCRIPTION:
Allogenic hematopoietic stem cell transplantation (allo-HSCT) is a curative, established treatment modality for a variety of malignant and nonmalignant hematologic disorders. Despite an increase in patient survival with HSCT, Graft-Versus-Host Disease (GVHD), in which donor immune cells detect recipient cells as foreign and attack the host tissue, is associated with significant morbidity and mortality after allo-HSCT. Ocular surface involvement is one of the most common manifestations of chronic GVHD with up to 60-90% of patients affected. Dry eye (DE) is the typical finding in ocular GVHD, and severe, chronic inflammation plays a crucial role in the pathogenesis. Therefore, topical steroids have been commonly used in patients with ocular GVHD (oGVHD). Although a healing effect of topical steroids has been shown in oGVHD, the efficacy of treatment might be reduced if it is not applied appropriately; poor patient compliance and improper drop administration (such as missing the eye and instilling an insufficient amount of medication) might diminish medication efficacy. Additionally, even if drops are applied appropriately, only approximately 5% of the administered dose can reach the target tissue because of blinking, nasolacrimal drainage, and low corneal permeability. Furthermore, the intermittent administration of topical drops results in a variable drug concentration in the target tissue and produces a suboptimal pharmacologic effect. Additionally, the prolonged use of topical steroids can also be toxic to the ocular surface due to preservatives such as benzalkonium chloride, which is used for its anti-microbial properties to prevent the contamination of drops. This toxicity might further disrupt the corneal epithelial barrier, which is already disrupted because of existing ocular surface inflammation.

To address all of these obstacles associated with topical steroids in patients with oGVHD, a sustained-released preservative-free intracanalicular insert (Dextenza, Ocular Therapeutix) may be beneficial. The purpose of this clinical trial is evaluate the safety and efficacy of Dextenza intracanalicular inserts in patients with ocular GVHD.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed as chronic ocular GVHD
* Age >= 18 years
* Corneal Fluorescein Staining ≥ 4
* Ocular Surface Disease Index ≥22.

Exclusion Criteria:

* History of immune diseases other than GVHD, herpetic keratitis or ocular malignancy
* Treatment regimen changes with topical cyclosporine, autologous serum, anakinra, or oral tetracycline compounds within 30 days prior to enrollment;
* Treatment regimen changes with systemic immunosuppressants or topical anti-glaucoma medications within 15 days prior to enrollment
* Current use of topical steroids more than twice a day
* Current or history of steroid induced ocular hypertension or glaucoma
* Family history of steroid induced ocular hypertension or glaucoma
* History of any intra-ocular surgery in the past 3 months or contact lens use within 2 weeks prior to enrollment
* History of collagen (prolong) intra-canalicular plug within 6 months
* Inability to cooperate for a comprehensive ocular examination
* History of lid deformity or neuroparalytic lid disease
* Active ocular infection including herpetic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-12-13 (Actual); Study Completion 2021-12-13 (Actual)

PRIMARY OUTCOMES:
Corneal Fluorescein Staining Score | 4 weeks
  Difference in the reduction of corneal fluorescein staining (CFS) compared to the contralateral eye. The cornea is divided into five zones (central, superior, temporal, nasal, and inferior) and for each zone, the severity of corneal fluorescein staining is graded on a scale from 0 to 3. Therefore, the maximum score is 15 for each eye. A higher score correlates to higher severity.
Lissamine green staining score | 4 Weeks
  The difference in the reduction of lissamine green staining compared to the contralateral eye. Six regions are graded for each eye (3 nasal conjunctival regions and 3 temporal conjunctival regions) from 0-3. Thus, a maximum score of 18 is possible for each eye. A higher score correlates to higher severity.
Symptomatic Relief | 4 Weeks
  The difference in symptomatic relief from baseline to 4 weeks, as compared to the contralateral eye using The Symptom Assessment Questionnaire iN Dry Eye Questionnaire (SANDE). SANDE is a visual analog scale questionnaire that quantifies the severity and frequency of dry eye symptoms. Subjects mark on a 100 mm horizontal linear visual analog scale, with a pen or pencil, their frequency, and severity. By measuring, in mm, where each scale was marked, a score can be obtained, from 0 to 100, where a higher score correlates to more frequent and more severe symptoms.

SECONDARY OUTCOMES:
The Symptom Assessment Questionnaire iN Dry Eye Questionnaire | 8 Weeks
  The difference in the improvement of the symptom assessment in dry eye (SANDE) questionnaire score compared to the contralateral eye at 4 and 8 week. SANDE is a visual analog scale questionnaire that quantifies the severity and frequency of dry eye symptoms. Subjects mark on a 100 mm horizontal linear visual analog scale, with a pen or pencil, their frequency, and severity. By measuring, in mm, where each scale was marked, a score can be obtained, from 0 to 100, where a higher score correlates to more frequent and more severe symptoms.
Schirmer's Test | 8 Weeks
  The differences in the improvement of Schirmer's test compared to the contralateral eye. Topical anesthetic is placed in the eye, and Schirmers test strips are placed in the temporal fornix of each eye. Patients are then instructed to close their eyes and after 5 minutes, the Schirmer strips are removed. The amount of wetting of each strip is read off of the strip and recorded. Values range from 0 to 35. Lower scores indicate lower tear production and greater ocular surface disease.
Tear Break Up Time | 8 Weeks
  The differences in the improvement of Tear Break Up Time (TBUT) compared to the contralateral eye. After instillation of fluorescein, the patient is asked to close their eyes, then open the eye and keep it open. The amount of time between opening the eye and visible disruption of the tear film is recorded in seconds. The same procedure is repeated for the fellow eye. Time can range from 0 seconds (instantaneous break up) to >10 seconds. Lower times indicate greater ocular surface disease.

CONTACTS AND LOCATIONS:
Locations (1):
- Mass Eye and Ear, Boston, Massachusetts, United States